CLINICAL TRIAL: NCT06993948
Title: Hyperdynamic Left Ventricular Ejection Fraction as a Predictor of Mortality in Intensive Care Unit Patients With Septic Shock
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa Saeed Mohamed Hedia, Assistant Lecturer of Anesthesia, Intensive Care and Pain Management Department, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Other Study IDs: MD 260/2022
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hyperdynamic; Left Ventricular Ejection Fraction; Mortality; Intensive Care Unit; Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic shock group: Patients underwent left ventricular ejection fraction (LVEF) assessment using two-dimensional echocardiography using visual estimation.
  Interventions: Device: Transthoracic echocardiography

INTERVENTIONS:
Device: Transthoracic echocardiography — Transthoracic echocardiography (TTE) was carried out. The assessment of left ventricular ejection fraction (LVEF) relied primarily on two-dimensional echocardiography using visual estimation.

SUMMARY:
The study aimed to evaluate the cause and prognosis of hyperdynamic left ventricular ejection fraction in critically ill patients with sepsis.

DETAILED DESCRIPTION:
Cardiovascular dysfunction is increasingly being recognized as a significant complication in sepsis, affecting patient outcomes.

Among the key parameters used to evaluate cardiac performance is the left ventricular ejection fraction (LVEF), typically assessed via transthoracic echocardiography (TTE).

LVEF has been extensively studied; most investigations into preserved ejection fraction tend to group all values ≥50% together, thereby overlooking the potential clinical implications of LVEF ≥70%, often referred to as hyperdynamic LVEF (HDLVEF).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Both sexes.
* Patients who were diagnosed with septic shock.

Exclusion Criteria:

- Patients with previously documented abnormal transthoracic echocardiography (TTE) findings, such as severe valvular disease, poor echocardiographic windows, patients admitted to cardiothoracic intensive care unit (ICU), and those not meeting sepsis criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study involved 235 patients admitted to the Intensive Care Unit (ICU) from August 2022 to July 2023.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Intensive care unit mortality | 28 days post-procedure
  Such patients are admitted to the intensive care unit (ICU), where a definitive diagnosis of sepsis is established using the Sequential Organ Failure Assessment (SOFA) score. This validated scoring system is widely recognized for its ability to predict mortality by evaluating dysfunction across six critical organ systems: respiratory, cardiovascular, hepatic, coagulation, renal, and neurological. The SOFA score is initially calculated upon ICU admission and is subsequently updated every 24 hours, using the most abnormal clinical or laboratory values recorded during the preceding day.

SECONDARY OUTCOMES:
Discharge against medical advice | 28 days post-procedure
  Discharge against medical advice was recorded.
Incidence of patients who choose to leave the intensive care unit | 28 days post-procedure
  Incidence of patients who choose to leave the intensive care unit against medical advice.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Hedia DSM, Mahmoud HO, AbdelFattah AM, AbdelSalam EH, Mahmoud OS. Hyperdynamic left ventricular ejection fraction as a predictor of mortality in intensive care unit patients with septic shock. Heart Lung. 2025 Nov 29;76:106-112. doi: 10.1016/j.hrtlng.2025.11.015. Online ahead of print. PMID 41319356